CLINICAL TRIAL: NCT06111378
Title: A Comparative Investigation of the Effects of OMEGA 3 Fatty Acids on Lactation
Brief Title: Effect of OMEGA 3 Fatty Acids on Lactation Period
Status: Completed | Type: Observational
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Hayrunnisa Yesil Sarsmaz, Asistant Prof., Celal Bayar University
Other Study IDs: MCBU_lactation
Record Dates: First submitted 2022-12-01; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2022-12

CONDITIONS: Lactation Induced
Keywords: lactation; omega 3 fatty acid; fish oil; flaxseed oil; walnut oil; breast cancer
MeSH Terms: conditions — Breast Feeding; Breast Neoplasms | interventions — Fish Oils; Linseed Oil

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — breast tissues cells
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group 1:: control group (n:7)
- Group 2:: fish oil group (n:7)
  Interventions: Dietary Supplement: fish oil
- Group 3:: linseed oil group (n:7)
  Interventions: Dietary Supplement: linseed oil
- Group 4:: walnut oil group (n:7)
  Interventions: Dietary Supplement: walnut oil
- Group 5:: sham group (non-lactating rats) (n:4)

INTERVENTIONS:
Dietary Supplement: fish oil — fish oil
  Groups: Group 2:
Dietary Supplement: linseed oil — linseed oil
  Groups: Group 3:
Dietary Supplement: walnut oil — walnut oil
  Groups: Group 4:

SUMMARY:
The World Health Organization (WHO) and the United Nations Children's Fund (UNICEF)

recommend that babies be exclusively breastfed for the first 6 months from birth. The composition of breast

milk is dynamic and may vary according to the content of maternal nutrition. Maternal nutrition, on the other

hand, determines the quality of breast milk necessary for the adequate growth and health of infants. For this

reason, the content of the maternal diet is important during the lactation period, which is the critical stage that

can affect the development of infants.

Omega 3 fatty acids are essential unsaturated fatty acids that are not synthesized by the human body and must be obtained through diet. The polyunsaturated fatty acids (PUFAs) most abundant in the diet are short-chain omega 3 alpha linolenic acid (ALA) and omega 6 linoleic acid (LA), which are mostly found in vegetable oils. ALA is a plant-derived omega 3 fatty acid found in flaxseed, walnut, canola and soybean oils. Eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) are found in marine sources such as seafood and fish oils. Today, the use of Omega 3 fatty acid supplements is increasing during the lactation period. However, consumption of omega 3 fatty acid sources during pregnancy or lactation is thought to be an important factor in preventing cancer risk. In our study, the investigators aimed to compare the maternal diet and the consumption of fish oil, flaxseed oil and walnut oil supplements during the lactation period, to compare the amount of prolactin and DHA in the milk composition and to compare the protective effects against breast cancer with cancer stem cell markers. For this study, 32 healthy Wistar pregnant rats, weighing 200-250 g, 8-10 weeks pregnant and not included in any experiments, will be used. Supplementary oils will be administered by oral gavage, considering the 0.5 g/kg body weight of the pregnant rats according to the groups they are assigned to, during the entire standard lactation period (day 21), considering the day of birth of the pregnant rats as the 0th day of lactation. Mother rats will be sacrificed under anesthesia at the end of the 21st day of lactation, mammary tissues will be taken into appropriate solutions and histopathological and immunohistochemical examinations will be performed. In addition, cardiac blood will be drawn and blood and tissue biochemical analyzes will be performed.

ELIGIBILITY:
Inclusion Criteria:

* healthy rats

Exclusion Criteria:

* patient rats
* rats that cannot be gavaged

Ages: 8 Weeks to 10 Weeks | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: pregnant rats unpregnant female rats
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-12-17 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Analysis of the Effects of OMEGA 3 Fatty Acids on Lactation | Baseline
  A Comparative Investigation of the maternal diet and the consumption of fish oil, flaxseed oil and walnut oil supplements during the lactation period. A Comparative Investigation of amount of prolactin and DHA in the milk composition and to compare the protective effects against breast cancer with cancer stem cell markers.

CONTACTS AND LOCATIONS:
Locations (1):
- Manisa Celal Bayar University, Yunusemre, Mani̇sa, Turkey (Türkiye)

REFERENCES:
- [Derived] Mutlu Durgut I, Yesil Sarsmaz H, Gurgen SG. A Comparative Study on the Effect of Omega-3 Fatty Acids on Lactation. Mol Nutr Food Res. 2026 Jan;70(2):e70393. doi: 10.1002/mnfr.70393. PMID 41572962